CLINICAL TRIAL: NCT03389555
Title: Ascorbic Ccid, Hydrocortisone, and Thiamine in Sepsis and Septic Shock - A Randomized, Double-Blind, Placebo-Controlled Trial
Brief Title: Ascorbic Acid, Corticosteroids, and Thiamine in Sepsis (ACTS) Trial
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Open Philanthropy (Other)
Responsible Party: Principal Investigator, Michael Donnino, Associate Professor of Emergency Medicine, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2017P000436
Record Dates: First submitted 2017-12-27; First posted 2018-01-03 (Actual); Results first posted 2021-01-29 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-01

CONDITIONS: Sepsis; Septic Shock; Metabolic Disturbance
Keywords: Sepsis; Metabolic Resuscitation
MeSH Terms: conditions — Sepsis; Shock, Septic | interventions — Ascorbic Acid; Thiamine; Hydrocortisone; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Vitamin C, Vitamin B1, Corticosteroids (Experimental): The combination of vitamin C, vitamin B1, hydrocortisone :
  * Vitamin C (ascorbic acid) 1.5g every 6 hours x 4-days
  * Vitamin B1 (thiamine) 100mg every 6 hours x 4-days
  * Hydrocortisone 50mg every 6 hours x 4-days
  Interventions: Drug: vitamin C, vitamin B1, hydrocortisone
- Placebo (Placebo Comparator): Normal Saline Solution (0.9%NaCl) in a volume to match all experimental arm components
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: vitamin C, vitamin B1, hydrocortisone — Vitamin C (1.5g) plus vitamin B1 (100mg) will be diluted in 100ml 0.9% NACL(normal saline) and administered IV every 6 hours for 4 days or until participant is discharged from the ICU. Hydrocortisone 50mg/ml will be administered via IV push over 1-2 minutes every 6hours for 4 days or until the patient is discharged from the ICU.
  Other Names: Ascorbic Acid; Thiamine
  Arms: Vitamin C, Vitamin B1, Corticosteroids
Drug: Normal saline — Normal saline (0.9% NaCl solution) volume to match all components
  Arms: Placebo

SUMMARY:
In this study, we aim to determine whether the combination of Ascorbic Acid (Vitamin C), Thiamine (Vitamin B1), and Corticosteroids improves the trajectory of organ failure and reduces mortality in patients with sepsis and septic shock as compared to placebo.

DETAILED DESCRIPTION:
Sepsis and Septic Shock are common and highly morbid clinical conditions without any specific therapy aside from antibiotics. A recent quasi-experimental study (Marik et. al., PMID 27940189) demonstrated a remarkable benefit when the combination of Ascorbic Acid (Vitamin C), Corticosteroids, and Thiamine (Vitamin B1) were given to patients with sepsis. In particular, patients who received this combination of medications required a shorter amount of time on vasopressors, suffered less organ failure, and had improved mortality. Vitamin C has long been suggested for treatment of patients with severe infection as it exerts significant anti-oxidant effects and reduces endothelial permeability. Corticosteroids, a mainstay of therapy for refractory shock in sepsis, have also been shown to enhance the beneficial cellular effects of vitamin C. Finally, thiamine has been shown to be an effective mitochondrial resuscitator in sepsis, especially for the ~30% of septic shock patients who present with thiamine deficiency (Donnino et. al, PMID 26771781).

In this study, we aim to reproduce the findings of Marik et. al. using a more rigorous study design (i.e. a blinded, randomized clinical trial) and focus on the important clinical outcomes of organ failure and death.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patient (age ≥ 18 years)
2. Suspected (cultures drawn and antibiotic given) or confirmed (via culture results) infection
3. Receiving vasopressor (norepinephrine, phenylephrine, epinephrine, dopamine, angiotensin II or vasopressin)

Exclusion Criteria:

1. Member of a protected population (pregnant, prisoner)
2. Known kidney stones within the past 1 year (except for asymptomatic, incidentally noted stones on imaging)
3. End stage renal disease (ESRD) requiring dialysis
4. Known Glucose-6-Phosphate Dehydrogenase deficiency
5. Known Hemachromatosis
6. Comfort Measures Only status
7. Anticipated death within 24-hours despite maximal therapy (as determined by the enrolling physician)
8. Receiving supplemental thiamine in a dose greater than that contained in a multivitamin
9. Clinical indication for steroids (e.g. chronic use) as determined by the clinical team providing this drug
10. Clinical indication for thiamine as determined by the clinical team providing this drug
11. Clinical indication for ascorbic acid as determined by the clinical team providing this drug
12. Known allergy to vitamin C, hydrocortisone, or thiamine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2018-02-09 (Actual); Primary Completion 2019-11-26 (Actual); Study Completion 2020-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael W Donnino, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (13):
- United States (13):
  - Mayo Clinic - Arizona, Phoenix, Arizona
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Mount Auburn Hospital, Cambridge, Massachusetts
  - Detroit Receiving Hospital, Detroit, Michigan
  - Harper University Hospital, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Sinai Grace Hospital, Detroit, Michigan
  - Beaumont Hospital, Royal Oak, Michigan
  - North Shore University Hospital, Manhasset, New York
  - Long Island Jewish Hospital, New York, New York
  - University Of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - The University of Texas Health Science Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Marik PE, Khangoora V, Rivera R, Hooper MH, Catravas J. Hydrocortisone, Vitamin C, and Thiamine for the Treatment of Severe Sepsis and Septic Shock: A Retrospective Before-After Study. Chest. 2017 Jun;151(6):1229-1238. doi: 10.1016/j.chest.2016.11.036. Epub 2016 Dec 6. PMID 27940189
- [Background] Moskowitz A, Andersen LW, Cocchi MN, Karlsson M, Patel PV, Donnino MW. Thiamine as a Renal Protective Agent in Septic Shock. A Secondary Analysis of a Randomized, Double-Blind, Placebo-controlled Trial. Ann Am Thorac Soc. 2017 May;14(5):737-741. doi: 10.1513/AnnalsATS.201608-656BC. PMID 28207287
- [Background] Donnino MW, Andersen LW, Chase M, Berg KM, Tidswell M, Giberson T, Wolfe R, Moskowitz A, Smithline H, Ngo L, Cocchi MN; Center for Resuscitation Science Research Group. Randomized, Double-Blind, Placebo-Controlled Trial of Thiamine as a Metabolic Resuscitator in Septic Shock: A Pilot Study. Crit Care Med. 2016 Feb;44(2):360-7. doi: 10.1097/CCM.0000000000001572. PMID 26771781
- [Derived] Grossestreuer AV, Moskowitz A, Andersen LW, Holmberg MJ, Konacki V, Berg KM, Chase M, Cocchi MN, Donnino MW. Effect of Ascorbic Acid, Corticosteroids, and Thiamine on Health-Related Quality of Life in Sepsis. Crit Care Explor. 2020 Nov 23;2(12):e0270. doi: 10.1097/CCE.0000000000000270. eCollection 2020 Dec. PMID 33251516
- [Derived] Moskowitz A, Huang DT, Hou PC, Gong J, Doshi PB, Grossestreuer AV, Andersen LW, Ngo L, Sherwin RL, Berg KM, Chase M, Cocchi MN, McCannon JB, Hershey M, Hilewitz A, Korotun M, Becker LB, Otero RM, Uduman J, Sen A, Donnino MW; ACTS Clinical Trial Investigators. Effect of Ascorbic Acid, Corticosteroids, and Thiamine on Organ Injury in Septic Shock: The ACTS Randomized Clinical Trial. JAMA. 2020 Aug 18;324(7):642-650. doi: 10.1001/jama.2020.11946. PMID 32809003
- [Derived] Moskowitz A, Yankama T, Andersen LW, Huang DT, Donnino MW, Grossestreuer AV; ACTS Clinical Trial Investigators. Ascorbic Acid, Corticosteroids and Thiamine in Sepsis (ACTS) protocol and statistical analysis plan: a prospective, multicentre, double-blind, randomised, placebo-controlled clinical trial. BMJ Open. 2019 Dec 17;9(12):e034406. doi: 10.1136/bmjopen-2019-034406. PMID 31852712

RESULTS

PARTICIPANT FLOW:
Groups:
- Vitamin C, Vitamin B1, Corticosteroids: The combination of vitamin C, vitamin B1, hydrocortisone :
  * Vitamin C (ascorbic acid) 1.5g every 6 hours x 4-days
  * Vitamin B1 (thiamine) 100mg every 6 hours x 4-days
  * Hydrocortisone 50mg every 6 hours x 4-days
  vitamin C, vitamin B1, hydrocortisone: Vitamin C (1.5g) plus vitamin B1 (100mg) will be diluted in 100ml 0.9%NACL and administered IV every 6 hours for 4 days or until participant is discharged from the ICU. Hydrocortisone 50mg/ml will be administered via IV push over 1-2 minutes every 6hours for 4 days or until the patient is discharged from the ICU.
Period: Overall Study
Arm/Group | Vitamin C, Vitamin B1, Corticosteroids | Placebo
Started | 103 | 102
Completed | 101 | 99
Not Completed | 2 | 3
Not completed — Protocol Violation | 1 | 3
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vitamin C, Vitamin B1, Corticosteroids | Placebo | Total
Number analyzed (Participants) | 101 | 99 | 200
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.9 (15.0) | 67.7 (13.9) | 68.2 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 45 | 89
  Male | 57 | 54 | 111
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Excluded 10 patients in intervention arm and 6 patients in placebo arm who did not have race data available.
  Participants
    White: number analyzed (Participants) | 91 | 93 | 184
    White | 68 | 73 | 141
    Black: number analyzed (Participants) | 91 | 93 | 184
    Black | 18 | 16 | 34
    Asian: number analyzed (Participants) | 91 | 93 | 184
    Asian | 5 | 3 | 8
    More than one Race: number analyzed (Participants) | 91 | 93 | 184
    More than one Race | 0 | 1 | 1
BMI, mean (SD) [Mean (Standard Deviation); unit: kg/m^2] | 28.8 (10.1) | 27.9 (8.4) | 28.3 (9.3)
Medical History, [Count of Participants; unit: Participants]
  # with Malignancy | 26 | 32 | 58
  # with Coronary Artery Disease | 26 | 26 | 52
  # with Congestive Heart Failure | 14 | 23 | 37
  Liver Disease | 11 | 7 | 18
Primary Infectious Source [Count of Participants; unit: Participants] — Population: Patients who did not have an identifiable primary infectious disease source were excluded from these tabulations (7 in intervention and 6 in placebo)
  Participants
    Pneumonia: number analyzed (Participants) | 94 | 93 | 187
    Pneumonia | 31 | 28 | 59
    Intra-abdominal: number analyzed (Participants) | 94 | 93 | 187
    Intra-abdominal | 30 | 23 | 53
    Urinary Tract Infection: number analyzed (Participants) | 94 | 93 | 187
    Urinary Tract Infection | 20 | 22 | 42
    Other: number analyzed (Participants) | 94 | 93 | 187
    Other | 13 | 20 | 33
Volume of Intravenous Fluids Prior to Study Drug [Median (Inter-Quartile Range); unit: mL] | 2000 [1062 to 3000] | 2000 [1125 to 3000] | 2000 [1093.5 to 3000]
Time from Vasopressor Initiation to First Study Drug [Median (Inter-Quartile Range); unit: hours] | 14.5 [8.1 to 19.1] | 13.0 [7.5 to 20.5] | 13.5 [8.0 to 19.8]
Time from Informed Consent to First Study Drug [Median (Inter-Quartile Range); unit: Hours] | 2.2 [1.7 to 3.0] | 2.0 [1.5 to 2.7] | 2.1 [1.6 to 2.9]
Baseline Cardiovascular Component of Total SOFA Score [Median (Inter-Quartile Range); unit: Units on a scale] — Baseline Cardiovascular Component of the Sequential Organ Failure Assessment (SOFA) score: The cardiovascular component of the SOFA score ranges from 0 (best) to 4 (worst), with a score of 0 indicating a mean arterial pressure of ≥ 70 mmHg, a score of 1 indicating a mean arterial pressure of < 70 mmHg, a score of 2 indicating dopamine dosing of ≤ 5 µg/kg/min or any dose of dobutamine, a score of 3 indicating norepinephrine dosing of ≤1mcg/kg/min (or equivalent) and a score of 4 indicating a norepinephrine dose >1mcg/kg/min (or equivalent).
  Units on a scale | 4 [3 to 4] | 4 [3 to 4] | 4 [3 to 4]
# on Mechanical Ventilation [Count of Participants; unit: Participants] | 48 | 44 | 92
# with Acute Respiratory Distress Syndrome [Count of Participants; unit: Participants] | 22 | 18 | 40
30 Day Predicted Survival [Count of Participants; unit: Participants] — At time of enrollment, the physician enrolling the patient is asked to predict the patient's chances of survival at the time-point 30 days after enrollment.
  Participants
    High Likelihood | 34 | 38 | 72
    Uncertain | 61 | 54 | 115
    Low Likelihood | 6 | 7 | 13
Lactate [Median (Inter-Quartile Range); unit: mmol/L] | 1.8 [1.3 to 2.9] | 1.8 [1.4 to 2.8] | 1.8 [1.3 to 2.8]

OUTCOME MEASURES:

1. Primary Outcome: Sequential Organ Failure Assessment (SOFA) Score at Baseline and 72 Hours
Description: Sequential Organ Failure Assessment (SOFA) Score at Baseline and 72 Hours. The SOFA score ranges from a minimum of 0 to a maximum of 24, with higher scores meaning worse outcomes.
Time Frame: Enrollment to 72-hours
Population: For the 72 hour SOFA score, patients who expired prior to that time point are excluded from the calculation of mean (SD) of the 72 hour SOFA score.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Vitamin C, Vitamin B1, Corticosteroids | Placebo
Number analyzed (Participants) | 101 | 99
Units on a scale
  Enrollment SOFA score | 9.1 (3.5) | 9.2 (3.2)
  72 hour SOFA score: number analyzed (Participants) | 90 | 88
  72 hour SOFA score | 4.4 (4.1) | 5.1 (4.3)
Statistical Analysis 1: Comparison: Vitamin C, Vitamin B1, Corticosteroids vs Placebo; The primary outcome was analyzed using a linear mixed-effects model where the correlation of within-patient repeated SOFA score measures was accounted for via the use of an unstructured variance-covariance matrix and linear contrasts. Covariates included age, sex, treatment group, time, and the interaction between treatment group and time. Study site was included as a random intercept. The model estimates the mean difference in SOFA score at 72 hours between treatment and control groups; Test type: Equivalence — Equivalence margin: if confidence interval for mean difference between SOFA scores at 72 hour time-point for two groups overlaps 0 (p-value > 0.05) scores considered to be equivalent. Note: The model estimates the mean difference in SOFA score at 72 hours between treatment and control groups, for those patient for whom a SOFA score could be calculated at the 72 hour time point (i.e patients that were alive at the 72 hour time point, 90 patients in the treatment and 88 patients in the control); p = 0.12, Mixed Models Analysis — A priori threshold for significance, p-value < 0.05; Mean Difference (Net) = -0.8, 95% CI 2-sided [-1.7 to 0.2]

2. Secondary Outcome: Renal Failure
Description: Development of renal failure as defined by a Kidney Disease Improving Global Outcomes [KDIGO] stage 3 or higher. There are 3 stages in the KDIGO scale with stage 3 being the worst (corresponds to renal failure).
  Stage 1- serum creatinine 1.5 to 1.9 times baseline OR an increase in serum creatinine ≥ 0.3 mg/dL OR urine output < 0.5ml/kg/hour for 6-12 hours. Stage 2- serum creatinine 2.0-2.9 times baseline OR urine output <0.5mg/kg/hour for ≥ 12 hours Stage 3- serum creatinine 3.0 times baseline (or serum creatinine of more than or equal to 4.0 mg/dl with an acute increase of at least 0.5 mg/dl) (OR) Urine output less than 0.3 ml/kg/hour for 24 hours or anuria for 12 hours or new renal replacement therapy
Time Frame: Enrollment until 7-days or discharge from the ICU
Measure: Count of Participants; unit: Participants
Arm/Group | Vitamin C, Vitamin B1, Corticosteroids | Placebo
Number analyzed (Participants) | 101 | 99
Participants | 32 | 27
Statistical Analysis 1: Comparison: Vitamin C, Vitamin B1, Corticosteroids vs Placebo; Logistic regression analysis evaluating the key secondary outcome of kidney failure in treatment group (intervention versus placebo) controlling for treatment site; Test type: Equivalence — For the key secondary outcome of kidney failure, 200 patients were estimated to provide 94% power, assuming that 30% of participants in the treatment group and 55% in the placebo group would develop kidney failure. If the adjusted risk difference from the logistic regression analysis overlaps 0, there was considered to be no difference between groups; p = 0.58, Regression, Logistic; Risk Difference (RD) = 3.0, 95% CI 2-sided [-10.0 to 20.0]

3. Secondary Outcome: 30-day Mortality
Description: Mortality rate
Time Frame: Enrollment until 30-days after enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Vitamin C, Vitamin B1, Corticosteroids | Placebo
Number analyzed (Participants) | 101 | 99
Participants | 35 | 29
Statistical Analysis 1: Comparison: Vitamin C, Vitamin B1, Corticosteroids vs Placebo; Cox Regression controlling for site used to identify hazard ratio for outcome of death for treatment versus intervention group. Null hypothesis is that hazard ratio is 1; Test type: Equivalence — If confidence interval for hazard ratio crosses 0, hazard of death assumed to be equivalent in the two groups; p = 0.05, Regression, Cox; Hazard Ratio (HR) = 1.3, 95% CI 2-sided [0.8 to 2.2]

4. Other Pre Specified Outcome: Ventilator Free Days
Description: Days not receiving invasive mechanical ventilation
Time Frame: Ventilator free days over the first 7-days after enrollment
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Vitamin C, Vitamin B1, Corticosteroids | Placebo
Number analyzed (Participants) | 101 | 99
Days | 6 [2 to 7] | 6 [0 to 7]
Statistical Analysis 1: Comparison: Vitamin C, Vitamin B1, Corticosteroids vs Placebo; Quantile regression controlling for site performed to compare treatment and control group's ventilator free days; Test type: Equivalence — If the confidence interval for the median difference in ventilator free days between groups crosses 0, the two groups are considered equivalent; p > 0.99, Quantile Regression; Median Difference (Net) = 0.0, 95% CI 2-sided [-1.9 to 1.9]

5. Other Pre Specified Outcome: Shock Free Days
Description: Days not receiving vasopressor
Time Frame: Vasopressor free days over the first 7-days after enrollment
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Vitamin C, Vitamin B1, Corticosteroids | Placebo
Number analyzed (Participants) | 101 | 99
Days | 5 [3 to 5] | 4 [1 to 5]
Statistical Analysis 1: Comparison: Vitamin C, Vitamin B1, Corticosteroids vs Placebo; Quantile regression controlling for site performed to compare treatment and control group's shock free days; Test type: Equivalence — If the confidence interval for the median difference in shock free days between groups crosses 0, the two groups are considered equivalent; p = 0.02, Quantile Regression; Median Difference (Net) = 1.0, 95% CI 2-sided [0.2 to 1.8]

6. Other Pre Specified Outcome: ICU Free Days
Description: Number of days that the patient was not in the ICU. Timeframe listed below.
Time Frame: From enrollment until 28 days after enrollment
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Vitamin C, Vitamin B1, Corticosteroids | Placebo
Number analyzed (Participants) | 101 | 99
Days | 22 [3 to 25] | 21 [4 to 25]
Statistical Analysis 1: Comparison: Vitamin C, Vitamin B1, Corticosteroids vs Placebo; Quantile regression controlling for site performed to compare treatment and control group's ICU free days; Test type: Equivalence — If the confidence interval for the median difference in ICU free days between groups crosses 0, the two groups are considered equivalent; p = 0.69, Quantile Regression; Median Difference (Net) = 1.0, 95% CI 2-sided [-3.0 to 6.0]

7. Other Pre Specified Outcome: Hospital Mortality
Description: Hospital mortality rate
Time Frame: Enrollment until hospital discharge, death, or 30-days. Whichever comes first.
Measure: Count of Participants; unit: Participants
Arm/Group | Vitamin C, Vitamin B1, Corticosteroids | Placebo
Number analyzed (Participants) | 101 | 99
Participants | 28 | 23
Statistical Analysis 1: Comparison: Vitamin C, Vitamin B1, Corticosteroids vs Placebo; Logistic regression analysis evaluating the key secondary outcome of hospital mortality in treatment group (intervention versus placebo) controlling for treatment site; Test type: Equivalence — If the adjusted risk difference from the logistic regression analysis overlaps 0, there was considered to be no difference between groups; p = 0.55, Regression, Logistic; Risk Difference (RD) = 3.0, 95% CI 2-sided [-10.0 to 20.0]

8. Other Pre Specified Outcome: Intensive Care Unit (ICU) Mortality
Description: ICU mortality rate
Time Frame: Enrollment until ICU discharge, death, or 30-days. Whichever comes first.
Measure: Count of Participants; unit: Participants
Arm/Group | Vitamin C, Vitamin B1, Corticosteroids | Placebo
Number analyzed (Participants) | 101 | 99
Participants | 23 | 20
Statistical Analysis 1: Comparison: Vitamin C, Vitamin B1, Corticosteroids vs Placebo; Logistic regression analysis evaluating the key secondary outcome of ICU mortality in treatment group (intervention versus placebo) controlling for treatment site; Test type: Equivalence — [test comment as in outcome 7, analysis 1]; p = 0.80, Regression, Logistic; Risk Difference (RD) = 2.0, 95% CI 2-sided [-10.0 to 10.0]

9. Other Pre Specified Outcome: Number of Participants With Delirium
Description: Describes if patient has delirium as defined by the Confusion Assessment Method (CAM)-ICU. The CAM-ICU method requires that the patient have 3 features to qualify for delirium:
  1. Acute Onset of Changes or Fluctuations in the Course of Mental Status (AND )
  2. Inattention (AND)
  3. Disorganized thinking (OR) Altered Level of Consciousness
Time Frame: On day 3 (at approximately 72 hours) after the first study drug dose
Population: We were able to assess CAM-ICU delirium on day 3 in only 83 patients from treatment and 76 patients from the control arm (unable to assess for remaining patients due to death or discharge)
Measure: Count of Participants; unit: Participants
Arm/Group | Vitamin C, Vitamin B1, Corticosteroids | Placebo
Number analyzed (Participants) | 83 | 76
Participants | 31 | 35
Statistical Analysis 1: Comparison: Vitamin C, Vitamin B1, Corticosteroids vs Placebo; Logistic regression analysis evaluating the key secondary outcome of occurrence of delirium in treatment group (intervention versus placebo) controlling for treatment site; Test type: Equivalence — [test comment as in outcome 7, analysis 1]; p = 0.16, Regression, Logistic; Risk Difference (RD) = -12, 95% CI 2-sided [-25 to 4]

10. Other Pre Specified Outcome: Hospital Disposition: Survivors Discharged Home
Description: Home hospital disposition in patients who survive to discharge
Time Frame: Enrollment until hospital discharge, death, or 30-days, whichever comes first.
Population: Population of patients who survived to hospital discharge. 73 patients in the treatment group and 76 patients in the control group survived to hospital discharge..
Measure: Count of Participants; unit: Participants
Arm/Group | Vitamin C, Vitamin B1, Corticosteroids | Placebo
Number analyzed (Participants) | 73 | 76
Participants | 34 | 35
Statistical Analysis 1: Comparison: Vitamin C, Vitamin B1, Corticosteroids vs Placebo; Logistic regression analysis evaluating home hospital disposition in survivors to hospital discharge in intervention versus placebo group controlling for treatment site; Test type: Equivalence — [test comment as in outcome 7, analysis 1]; p = 0.82, Regression, Logistic; Risk Difference (RD) = -1.8, 95% CI 2-sided [-18 to 14]

ADVERSE EVENTS:
Time Frame: Time from enrollment to hospital discharge, an average of 13.5 days for all patients
Arm/Group | Vitamin C, Vitamin B1, Corticosteroids | Placebo
All-Cause Mortality (participants affected / at risk) | 35/101 | 29/99
Serious Adverse Events (participants affected / at risk) | 13/101 | 12/99
Other Adverse Events (participants affected / at risk) | 0/101 | 0/99
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vitamin C, Vitamin B1, Corticosteroids (N=101) | Placebo (N=99)
Hyperglycemia (Endocrine disorders) | 12 (101) | 7 (99)
Hypernatremia (Metabolism and nutrition disorders) | 11 (101) | 7 (99)
New Hospital Acquired Infection (Infections and infestations) | 13 (101) | 12 (99)

LIMITATIONS AND CAVEATS:
Ongoing or planned corticosteroid use was the most common exclusion criterion, perhaps eliminating a subset of patients more likely to benefit from corticosteroids. Some patients were discharged alive from the ICU within 96 hours of enrollment; thus, many patients did not receive a full 4 days of study drug

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-12-13): https://cdn.clinicaltrials.gov/large-docs/55/NCT03389555/Prot_001.pdf
  • Statistical Analysis Plan (2018-12-13): https://cdn.clinicaltrials.gov/large-docs/55/NCT03389555/SAP_003.pdf